CLINICAL TRIAL: NCT02124382
Title: Living Donor Liver Transplantation in Children: Surgical and Immunological Results in 250 Recipients at Université Catholique de Louvain.
Brief Title: Living Donor Liver Transplantation in Children
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: CHIRPEDMG2012
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Pediatric Liver Transplanted Recipients; Healthy Donors
Keywords: liver failure; liver malignancy; metabolic diseases; Pediatric liver transplanted recipients and their healthy donors
MeSH Terms: conditions — Liver Failure; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the outcome of pediatric living donor liver transplantation (LDLT) regarding portal vein reconstruction, ABO-compatibility and impact of maternal donation on graft acceptance.

DETAILED DESCRIPTION:
Data from 250 pediatric LDLT recipients (and their donors), transplanted at Cliniques universitaires Saint-Luc between July 1993 and June 2012, were collected retrospectively using electronic data files. Results were analysed according to ABO matching and portal vein complications. Uni- and multi-variate analysis was used to study the impact of immunosuppression, gender match and maternal donation on acute rejection rate.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving a living donor liver transplant
* Adult living donors

Exclusion Criteria:

* No one

Max Age: 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 250 pediatric living donor liver transplant recipients 250 corresponding adult living donors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Patient and graft survival | 10 years
  Kaplan-Meier

SECONDARY OUTCOMES:
Portal vein complications | 10 years

OTHER OUTCOMES:
Graft rejection free survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Reding, Md-PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain